CLINICAL TRIAL: NCT06631287
Title: Randomized Double-Blind Placebo-Controlled Trial EValuating Baricitinib on PERSistent NEurologic and Cardiopulmonary Symptoms of Long COVID (REVERSE-LC)
Brief Title: Randomized Double-Blind Placebo-Controlled Trial EValuating Baricitinib on PERSistent NEurologic and Cardiopulmonary Symptoms of Long COVID
Acronym: REVERSE-LC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wes Ely (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Wes Ely, Professor, Allergy, Pulmonary, and Critical Care Medicine, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REVERSE-LC; R01AG085873 (NIH)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Long COVID; Sars-CoV-2 Infection; Coronavirus Infections; COVID-19
Keywords: COVID-19; Long COVID Drug Treatment; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Coronavirus Infections | interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: Investigators will use adequate allocation concealment using a computer-generated, permuted-block randomization with varying block size. Randomization (1:1) will be stratified by site, SARS CoV-2 confirmatory test (cohort 1), and opting into the LP sub-study. The block size and treatment allocation will only be known to a biostatistician creating the randomization list and the study pharmacist and will not be shared with trial investigators or any other study personnel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baricitinib (Experimental): Janus kinase inhibitor
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Baricitinib — 4mg encapsulated, pre-formed tablet PO once daily for 24 weeks.
  Other Names: OLUMIANT
  Arms: Baricitinib
Other: Placebo — Matched placebo capsule, PO once daily for 24 weeks.
  Arms: Placebo

SUMMARY:
The overarching goal of this study is to determine if baricitinib, as compared to placebo, will improve neurocognitive function, along with measures of physical function, quality of life, post-exertional malaise, effect of breathlessness on daily activities, post-COVID-19 symptom burden, and biomarkers of inflammation and viral measures, in participants with Long COVID.

DETAILED DESCRIPTION:
Since the emergence of the severe acute respiratory syndrome coronavirus 2 pathogen in late 2019, there have been over 680 million cases worldwide and over 6 million deaths. In the United States alone, there have been over 100 million cases and over 1 million deaths. Both novel vaccines and effective therapeutics have helped reduce mortality in well-resourced countries. Despite these advances, millions of patients subsequently experience a devastating post-acute infection syndrome known as post-acute sequelae of SARS-CoV-2 infection (PASC), or better known by patients as Long COVID (LC). In the United States alone, it is estimated that up to 18 million adults suffer from LC with persistent neurocognitive impairments (NCI) and cardiopulmonary symptoms such as dyspnea and exercise intolerance for months to years after acute COVID-19. Additionally, up to 1 in 5 patients who were working prior to contracting SARS-CoV-2 may not return to the workforce due to cognitive and physical impairments. The public health burden of LC is estimated to be the largest seen from an emerging disease in the last 100 years, yet there are currently no effective interventions.

These clear and objective changes in cognitive function and brain structure highlight the devastating and long-lasting effects of SARS-CoV-2 infection on survivors' long-term health, highlighting the need for effective therapies to improve long-term cognitive outcomes.

In addition to the devastating NCI that patients with LC experience, many survivors go on to experience activity-limiting dyspnea on exertion, exercise intolerance, and reduced physical function. In fact, patients who have not fully recovered physically 5 months after infection may fail to recover further by one year. Patients with LC experience significant self-reported physical symptoms including persistent fatigue and dyspnea as well as objective impairments in exercise capacity and physical function upon performance testing. These impairments, in addition to cognitive function and mental health, lead to significant reductions in quality of life for these survivors.

While viral reservoirs, systemic and organ-level inflammation are leading hypotheses for the mechanistic underpinnings of LC, no trials to date have investigated the use of agents targeting these mechanisms. Similar chronic inflammation plays a crucial role in the increased risk of cardiovascular disease (CVD) and NCI for people with HIV (PWH) as indicated by elevated soluble and cellular markers of inflammation, endothelial dysfunction, and hypercoagulability in this population. Activation of the Janus kinase (JAK)-STAT pathway, which drives a proinflammatory milieu, has been reported during HIV infection and is associated with CVD, NCI, and HIV persistence. Even in the absence of a viral infection, these same conditions and comorbidities are driven by a very similar chronic inflammatory state.

ELIGIBILITY:
INCLUSION CRITERIA:

In order to be eligible to participate in this investigation, an individual must meet all of the following criteria:

Cohort #1 (n=500):

1. Evidence of personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study and was willing and able to consent to participation.
2. Age ≥18 years old.
3. Documented SARS-CoV-2 infection 6 or more months prior to screening, confirmed with acceptable documentation that includes (at minimum) their name, the date the test was taken (must be after January 2020), and details specifying that the positive test was for SARS-CoV-2 infection.
4. Clinical evidence of Long COVID, as confirmed by the investigator's assessment:

   a. At least one symptom (listed below) that is new or worsened since the time of SARS-CoV-2 infection, not known to be attributable to another cause upon assessment by the study clinicians (MD, DO, NP, PA, RN, or equivalent).

   i. Systemic symptoms (e.g., fatigue, chills, post-exertional malaise), neurocognitive symptoms (e.g., trouble with memory/concentration ("brain fog"), headache, dysautonomia/postural orthostatic tachycardia syndrome, dizziness, unsteadiness, neuropathy, sleep disturbance), cardiopulmonary symptoms (e.g., chest pain, palpitations, shortness of breath, cough, fainting spells), musculoskeletal symptoms (e.g., muscle aches, joint pain), gastrointestinal symptoms (e.g., nausea, diarrhea). Although other symptoms (e.g., skin rash, hair loss, mental health symptoms, trouble with smell/taste, genitourinary symptoms) will be recorded and tracked, at least one core symptoms listed above must be present.

   b. Symptoms must be present for at least 6 months prior to screening. Symptoms that wax and wane must have been initially present at least 6 months prior to screening.

   c. Symptoms must be reported to have an impact on quality of life and/or everyday functioning and to be at least somewhat bothersome.

   d. Cognitive impairment present defined by having at least 20% positive items (answered subjectively worse or much worse) on the 41-item modified ECog questionnaire.

Cohort #2 (n=50):

1. Evidence of personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study and was willing and able to consent to participation.
2. Age ≥18 years old.
3. Clinical diagnosis of COVID infection between January 2020 and September 1, 2021 (i.e., before home tests were widely available).

   a. Clinical Criteria (Based on Council of State and Territorial Epidemiologists Standardized Surveillance Case Definition for COVID-19): i. At least two of the following symptoms: Fever (measured or subjective), chills, rigors, myalgia, headache, sore throat, new olfactory and taste disorder(s).

   -OR- ii. At least one of the following symptoms: Cough, shortness of breath, or difficulty breathing.

   -OR- iii. Severe respiratory illness with at least one of the following: clinical or radiographic evidence of pneumonia or Acute Respiratory Distress Syndrome (ARDS).

   -AND- iv. No alternate more likely diagnosis
4. Clinical evidence of Long COVID, as confirmed by the clinician's assessment:

   a. At least one symptom (listed below) that is new or worsened since the time of SARS-CoV-2 infection, not known to be attributable to another cause upon assessment by the study clinicians (MD, DO, NP, PA, RN, or equivalent).

   i. Systemic symptoms (e.g., fatigue, chills, post-exertional malaise), neurocognitive symptoms (e.g., trouble with memory/concentration ("brain fog"), headache, dysautonomia/postural orthostatic tachycardia syndrome, dizziness, unsteadiness, neuropathy, sleep disturbance), cardiopulmonary symptoms (e.g., chest pain, palpitations, shortness of breath, cough, fainting spells), musculoskeletal symptoms (e.g., muscle aches, joint pain), gastrointestinal symptoms (e.g., nausea, diarrhea). Although other symptoms (e.g., skin rash, hair loss, mental health symptoms, trouble with smell/taste, genitourinary symptoms) will be recorded and tracked, at least one core symptoms listed above must be present.

   b. Symptoms must be present for at least 6 months prior to screening. Symptoms that wax and wane must have been initially present at least 6 months prior to screening.

   c. Symptoms must be reported to have an impact on quality of life and/or everyday functioning and to be at least somewhat bothersome.

   d. Cognitive impairment present defined by having at least 20% positive items (answered subjectively worse or much worse) on the 41-item modified ECog questionnaire.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this investigation:

1. Qualifying Long COVID symptoms cannot be explained by an infection-associated chronic condition diagnosed prior to the onset of Long COVID (e.g., ME/CFS or other infection-associated chronic condition).
2. Pre-existing cognitive impairment not exacerbated by COVID-19, including but not limited to syphilis, as determined by study clinicians (MD, DO, NP, PA, RN, or equivalent), which may include a review of participant's history and medical records.
3. Severe cognitive, physical, or psychological disability preventing participation in the study, as determined by the investigator.
4. Moderate or High risk of suicidality, as determined by the modified Columbia Suicide Severity Rating Scale (mC-SSRS).
5. History of a major adverse cardiovascular event (MACE) within the 3 months prior to enrollment.
6. Current use of baricitinib or other disease-modifying antirheumatic drug (DMARDs); however, DMARDs with minimal immunomodulatory effects (hydroxychloroquine, i.e., Plaquenil, steroids used for less than 2 weeks, minocycline), are not exclusionary.
7. Known prior allergic reactions to components of the baricitinib.
8. Previously randomized in this study or in the last 30 days have been in another study investigating baricitinib.
9. Positive SARS-CoV-2 NAAT or rapid Antigen test in the 14 days prior to screening.
10. Venous thromboembolism in the past 6 months prior to screening or felt to be at increased risk of thrombosis by the investigator.
11. Malignancy or lymphoproliferative disorder not in remission for at least 5 years. Local non-melanoma skin cancers that are definitively managed are not exclusionary.
12. Previous admission to an ICU for treatment of acute COVID-19 infection.
13. Estimated glomerular filtration rate of < 30 mL/min/1.73m2, as calculated using the CKD-EPI 2021 equation.
14. Absolute Neutrophil Count (ANC) <1000 cells/mm3, confirmed on repeat testing.
15. Absolute Leukocyte Count (ALC) <100 cells/mm3.
16. Evidence of severe liver disease at the time of screening, defined as Bilirubin > 1.5 X ULN or AST or ALT > 2x ULN.
17. Alkaline Phosphatase (ALP) ≥ 3x ULN.
18. Creatine Phosphokinase (CPK) ≥ 3x ULN.
19. Hemoglobin (HgB) < 8 g/dL, confirmed on repeat testing.
20. Platelets <100,000 cells/mm3, confirmed on repeat testing.
21. Platelets >500,000 cells/mm3, confirmed on repeat testing.
22. Total fasting cholesterol ≥ 280 mg/dL, confirmed on repeat testing.
23. Fasting LDL ≥ 180 mg/dL, confirmed on repeat testing.
24. Positive Hepatitis B surface antigen or Hepatitis B core antibody. Note: Individuals with a positive Hepatitis B core antibody will be excluded even in the presence of a positive Hepatitis B surface antibody due to the risk of reactivation.
25. Positive for Hepatitis C at the time of Screening. Note: treated or cleared Hepatitis C is not exclusionary.
26. Symptomatic herpes zoster infection (i.e., visible herpetic skin lesions of Zoster) within 3 months prior to study screening, or any history of disseminated/complicated herpes zoster or herpes simplex infection (e.g., VZV encephalitis).
27. History of untreated latent tuberculosis infection (diagnosed with QuantiFERON-TB Gold Plus testing) or active tuberculosis whether treated or untreated. Note: those with a positive PPD who have a history of BCG vaccine and a negative QuantiFERON-TB Gold Plus test will remain eligible).
28. History of current or recent (< 30 days from screening) sepsis or clinically significant viral, bacterial, fungal, or parasitic infection, according to the determination of the investigator.
29. Participants with HIV will be excluded if they have been on ART <1 year, have a CD4+ T cell count <500 cells/ml (confirmed on repeat), or have two consecutive HIV plasma RNA viral load > 48 copies/mL within 1 year of study screening, including requiring the most recent within 3 months of screening. Blips (VL > 48 copies/mL but < 200 copies/mL) are permitted if preceded and followed by values below the assay limit of quantification.
30. Immunocompromised as defined by NIH COVID-19 guidelines (see Appendix) and, in the opinion of the investigator, at an unacceptable risk for participating in the study.
31. Treatment with another investigational drug or device as part of an interventional study within 30 days of study screening.
32. In the opinion of the investigator, unable to reliably follow-up for the duration of the study and/or are unable to follow study restrictions/procedures.
33. Persons of childbearing potential under age 55 who are unwilling or unable to abstain from sex or to use at least one acceptable method of contraception from the time of screening though at least 28 days after the end of the study intervention period. Note: Acceptable methods include barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUDs), other contraceptives, oral contraceptive pills, and surgical sterilization. Participants unwilling to be counseled about risks related to pregnancy or breastfeeding.
34. Currently pregnant or breastfeeding or planning to become pregnant or breastfeed during the course of the study.
35. Participants actively breastfeeding, who are unwilling to stop breastfeeding for the duration of the trial.
36. Currently incarcerated

NOTE RE: History of major adverse cardiovascular event (MACE) or traditional risk factors including smoking. For REVERSE-LC, MACE is defined as acute myocardial infarction and stroke. The study team will discuss the risks and benefits of baricitinib and CV events with the participant prior to study entry.

NOTE RE: EBV/CMV Seropositivity - The investigators will not exclude participants based on EBV or CMV seropositivity. The investigators already know that serologic evidence suggesting recent EBV reactivation is associated with Long COVID fatigue and high level EBV responses are associated with neurocognitive Long COVID, but that EBV viremia and IgM is rare. The investigators believe there is equipoise with regard to the potential effects of baricitinib on EBV - it is as likely that inflammation drives EBV reactivation, just as EBV can drive inflammation. For this reason, the investigators think this is best studied as a biological factor correlated with outcomes and that the investigators should not deliberately include or exclude people based on this. CMV seropositivity is associated with improved Long COVID outcomes. Results are not required for screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
CNS-Vital Signs Global Cognitive Index | Month 6
  Objective neuropsychological function determined using the CNS-Vital Signs Global Cognitive Index between study arms at 6-months, adjusted for baseline.
  CNS-Vital Signs Global Cognitive Index subscale is an average score derived from the domain scores or a general assessment of the overall neurocognitive status of the participant. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.

SECONDARY OUTCOMES:
Objective neuropsychological function domains of executive function, memory, processing speed, and motor speed including the CNS-Vital Signs subscale tests at 6-months. | Month 6
  CNS-Vital Signs Global Cognitive Index is an average score derived from the domain scores or a general assessment of the overall neurocognitive status of the participant. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Objective neuropsychological function domains of executive function, memory, processing speed, and motor speed including the CNS-Vital Signs subscale tests at 12-months. | Month 12
  CNS-Vital Signs Global Cognitive Index subscale is an average score derived from the domain scores or a general assessment of the overall neurocognitive status of the participant. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Modified Everyday Cognition (mECog) | Months 3, 6 and 12
  Subjective participant-reported cognitive impairment including modified Everyday Cognition (mECog) scale at 3-, 6-, and 12-months.
  The mECog measure uses the sum score of all of the subscales, and the items are reverse coded (i.e., 1= "Better or no change", 2="Questionable/occasionally worse", 3="Consistently a little worse", 4="Consistently much worse"), meaning that lower scores are better. Reported total scores range from 39 (Better or no change) to 156 (Consistently much worse).
Exercise capacity including the 6-minute walk test (6MWT) at 6- and 12-months | Months 6 and 12
  Total distance in meters walked in 6 minutes
Cardiopulmonary exercise testing (CPET) | Months 6 and 12
  Cardiorespiratory fitness (peak VO2) using cardiopulmonary exercise testing (CPET) at 6- and 12- months. CPET is used to assess change in exercise tolerance as measured by VO2max.
Quality-of-life measures including the EuroQOL-5D-5L at 3-, 6-, and 12-months | Months 3, 6, and 12
  The 5-Level EuroQol-5D health questionnaire (EQ-5D-5L) is a standardized instrument for use as a measure of health outcome that includes a descriptive system consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The index value total (which is country-specific) ranges from a minimum value of -1 to a maximum value of +1. A higher EQ-5D-5L index value represents better quality of life (QoL), thus a positive change in the index value represents improved QoL.
Post-exertional malaise including the modified De Paul Symptom Questionnaire - Post-Exertional Malaise (mDSQ-PEM) at 6- and 12-months | Months 6 and 12
  The mDSQ-PEM has 10 questions (5 on severity and 5 on frequency) scored 0-4, with higher scores indicating greater post exertional malaise severity.
Effect of breathlessness on daily activities including the Modified Medical Research Council Dyspnea Scale (mMRC) at 6- and 12-months | Months 6 and 12
  Modified Medical Research Council Dyspnea Scale (mMRC) ranges from grade 0 to 4. 0 means no dyspnea, 1 means mild dyspnea (respiratory distress when moving quickly and climbing slightly uphill); 2 means moderate dyspnea (walking slower than peers when walking straight on, stopping to breathe); 3 means severe dyspnea (stopping to breathe after walking about 100 m or for a few minutes) and 4 means very severe dyspnea (getting out of breath while doing daily chores at home, while putting on and taking off clothes and while going to toilet).
Post COVID-19 symptom burden including the Symptom Burden Questionnaire for Long COVID (SBQ-LC) Circulation Subscale at 1-, 3-, 6-, and 12-months | Months 1, 3, 6, and 12
  The SBQ-LC Circulation Subscale consists of 5 questions with a score of 0-11 where higher scores indicate greater circulation-related symptom burden.
General participant-reported outcomes using the PROMIS-29 at 1-, 3-, 6-, and 12-months | Months 1, 3, 6, and 12
  The Patient-Reported Outcomes Measurement Information System (PROMIS)-29 has 29 questions across seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) each scored 1-5, with higher scores indicating worse symptoms or better function, depending on the domain.
Cognitive participant-reported outcomes using the PROMIS-Cognitive Function-Short Form 8a at 1-, 3-, 6-, and 12-months | Months 1, 3, 6, and 12
  The Patient-Reported Outcomes Measurement Information System-Cognitive Function-Short Form 8a (PROMIS-CF-8a) has 8 questions, each scored 1-5, with higher scores indicating better cognitive function.
Mental health measures including depression, anxiety, and stress using the DASS-21 at 6- and 12-months | Months 6 and 12
  The Depression Anxiety Stress Scale (DASS)-21 is a set of three (depression, anxiety, stress) self reported scales. Depression: Normal 0-9, Mild 10-13, Moderate 14-20, Severe 21-27, Extremely Severe 28+. Anxiety Normal 0-7, Mild 8-9, Moderate 10-14, Severe 15-19, Extremely Severe 20+. Stress Normal 0-14, Mild 15-18, Moderate 19-25, Severe 26-33, Extremely Severe 34+.
Orthostatic intolerance using the Orthostatic Intolerance Questionnaire (OIQ) at 3-, 6-, and 12-months | Months 3, 6, and 12
  Each subscale is scored on a 0-10 scale, with higher scores reflecting more severe symptoms compared to few/no symptoms at lower scores. The OISA has a total possible score of 40 and the OIDAS a total possible score of 60.
Autonomic dysfunction using the COMPASS-31 at 3-, 6-, and 12-months. | Months 3, 6, and 12
  The Composite Autonomic Symptom Score (COMPASS)-31 has 31 questions across six health domains (orthostatic Intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor), scored 0-4 with higher scores indicating greater autonomic symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Wes Ely, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - University of Minnesota, Minneapolis, Minnesota
  - Vanderbilt University Medical, Nashville, Tennessee